CLINICAL TRIAL: NCT04882176
Title: A Phase I/II, First-in-Human, Open-Label, Dose-Escalation and Dose-Extension Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Efficacy of LM-061 Tablet in Subjects With Advanced Tumours
Brief Title: A Clinical Study Preliminary Efficacy of LM-061 Tablet in Subjects With Advanced Tumours
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Not meeting expected endpoints
Sponsor: LaNova Medicines Limited (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LM061-01-101
Record Dates: First submitted 2021-04-22; First posted 2021-05-11 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2021-04

CONDITIONS: Advanced Tumours

STUDY DESIGN:
Intervention Model Description: Arm1: LM-061 2.5mg P.O QD Arm2: LM-061 5mg, P.O QD Arm3: LM-061 10mg, P.O QD Arm4: LM-061 20mg, P.O QD Arm5: LM-061 30mg, P.O QD Arm6: LM-061 40mg, P.O QD Arm7: LM-061 60mg, P.O QD
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (7):
- LM061 Dose Escalation Level 1, 2.5mg (Experimental): The dose escalation scheme using the the accelerated titration design for dose 1 and the i3+3 design for the remaining doses.
  first dose: 2.5mg QD, n=1;
  Interventions: Drug: LM-061
- LM061 Dose Escalation Level 2, 5mg (Experimental): The dose escalation scheme using the the accelerated titration design for dose 1 and the i3+3 design for the remaining doses.
  second dose: 5mg QD, n=3;
  Interventions: Drug: LM-061
- LM061 Dose Escalation Level 3, 10mg (Experimental): The dose escalation scheme using the the accelerated titration design for dose 1 and the i3+3 design for the remaining doses.
  third dose: 10mg QD, n=3;
  Interventions: Drug: LM-061
- LM061 Dose Escalation Level 4, 20mg (Experimental): The dose escalation scheme using the the accelerated titration design for dose 1 and the i3+3 design for the remaining doses.
  fourth dose: 20mg, n=3;
  Interventions: Drug: LM-061
- LM061 Dose Escalation Level 5, 30mg (Experimental): The dose escalation scheme using the the accelerated titration design for dose 1 and the i3+3 design for the remaining doses.
  fifth dose: 30mg, n=3;
  Interventions: Drug: LM-061
- LM061 Dose Escalation Level 6, 40mg (Experimental): The dose escalation scheme using the the accelerated titration design for dose 1 and the i3+3 design for the remaining doses.
  sixth dose: 40mg, n=9;
  Interventions: Drug: LM-061
- LM061 Dose Escalation Level 7, 60mg (Experimental): The dose escalation scheme using the the accelerated titration design for dose 1 and the i3+3 design for the remaining doses.
  seventh dose: 60mg, n=15;
  Interventions: Drug: LM-061

INTERVENTIONS:
Drug: LM-061 — The subjects in each dose level will be administered single oral dose of LM-061 tablet on C0D1, and washout for 5 days. After that, the subjects will be administered multiple oral doses once daily (QD) in continuous 28 days (4 weeks) per treatment cycle, until meet the treatment termination criteria, including disease progression or unaccepted toxicity, etc. After obtaining MTD/RP2D, the Safety Review Committee (SRC) may combine the data of safety, PK, and preliminary efficacy to explore other dosing schedules (such as 3 weeks on and 1 week off).
  Other Names: Kinase inhibitor

SUMMARY:
This is a phase I/II, open-label, dose escalation and dose extension study to evaluate the safety, tolerability, PK, and preliminary efficacy of LM-061 in subjects with advanced tumors.

DETAILED DESCRIPTION:
This is a phase I/II, open-label, dose escalation and dose extension study to evaluate the safety, tolerability, PK, and preliminary efficacy of LM-061 in subjects with advanced tumors.

The study schedule includes screening visit (28 days prior to accept the investigational medicinal product (IMP)), treatment visit (accept IMP for the first time to the end of treatment (EOT)/early withdrawal), and follow-up visit (28 days after the EOT/early withdrawal).

ELIGIBILITY:
Inclusion Criteria:

* Volunteer to participate in clinical study, sign a written informed consent form, and be able to comply with clinical visits and study related procedures;
* Male or female subjects 18 to 75 years old (both inclusive) when sign the informed consent;
* Study population;
* Dose Escalation the subjects with advanced malignant tumors confirmed by histology or cytology, and have failed standard treatment, or have no standard treatment, or not suitable for standard treatment at present;
* Dose Extension patients with advanced solid tumors with abnormal c-Met, including EGFR-TKI-resistant non-small cell lung cancer and pulmonary sarcomatoid adenocarcinoma, diagnosed histologically or cytologically, who have failed standard therapy, or who do not have standard treatment regimens, or who are not suitable for standard therapy at this stage;Papillary renal cell carcinoma;Metastatic or locally advanced unresectable gastric adenocarcinoma with at least first-line standard treatment;
* ECOG score 0-1;
* C-MET abnormalities are defined by central laboratory as the situation that meets one of the following: Abnormal expression of c-Met immunohistochemistry (IHC) : strong staining (2+ or above) in more than 50% of tumor cells; MET amplification positive: MET/CEP 7 ≥2 or GCN ≥5; MET exon14-skipping mutation;
* The estimated survival time is not less than 3 months;
* The functional of bone marrow reserve and organs must meet the following requirements (without ongoing continuous supportive treatment): Bone marrow reserve: Neutrophil count (NE#) ≥ 1.5×109/L, platelet count (PLT) ≥90 ×109/L; hemoglobin (HGB) > 9.0 g/dL (no blood transfusion or hematopoietic stimulating factor therapy within 14 days); Coagulation function: activated partial thromboplastin time (APTT) prolong ≤ 1.5× upper limit of normal (ULN), and international standard ratio (INR) ≤ 1.5; Liver function: total bilirubin (TBIL) ≤ 1.5×ULN, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5×ULN (if there is liver metastasis, ALT or AST≤ 5×ULN); Kidney function: Creatinine clearance rate ≥50 mL/min (using Cockcroft-Gault formula, see Appendix 1) or serum creatinine ≤1.5×ULN; qualitative urine protein ≤1+ or qualitative urine protein ≥2+, but 24-hour urine protein <1g; Cardiac function: left ventricular ejection fraction (LVEF) ≥ 50%; ECG is basically normal, and corrected QT interval (QTcF) ≤450 ms and 470 ms for male and female, respectively;
* According to RECIST v1.1 criteria, there should be at least one evaluable tumor focus in the dose escalation phase;At least one measurable tumor was present during the dose expansion phase;
* Eligible subjects with fertility (male and female) must agree to use reliable contraceptive methods (hormonal or barrier method or abstinence, etc.) with their partners during the trial period and at least 3 months after the last administration; women of childbearing age (Refer to Appendix 2 for definitions) The subject's serum pregnancy test must be negative within 7 days prior to the first administration.

Exclusion Criteria:

* Have received chemotherapy, radiotherapy, biological therapy, endocrine therapy, immune checkpoint inhibitor therapy and other anti-tumour treatments within 4 weeks prior to first dose of IMP, except for the following items:
* Subjects was diagnosed as acute promyelocytic leukemia (APL), breakpoint cluster region-abelson (BCR-ABL)-positive leukemia (i.e., chronic myelogenous leukemia in blast crisis), active central nervous system leukemia, or AML secondary to prior chemotherapy for other neoplasms;
* Have used nitrosourea or Mitomycin C within 6 weeks prior to first dose of IMP;
* Have used oral fluorouracil and small molecule targeted drugs within 2 weeks or 5 half-lives of the drugs prior to first dose of IMP (whichever is longer);
* Have received other unmarketed clinical study drugs or treatments within 4 weeks prior to first dose of IMP;
* Have undergone major organ surgery (excluding biopsy) or have had significant trauma or invasive dental procedures (such as tooth extraction, dental implant) within 4 weeks prior to first dose of IMP, or required elective surgery during the study period;
* Have serious unhealable wounds/ulcers/bone fractures within 4 weeks prior to first dose of IMP;
* Are taking (or cannot be stopped at least 1 week prior to first dose of IMP) any drug that is known to strongly inhibit or induce CYP3A4 (see Appendix 5 for details);
* The histopathological type of the tumour is head and neck or lung squamous cell carcinoma, or other tumours with bleeding tendency as judged by the investigator;
* Bleeding events of grade 3 or above occurred within 6 months before the first dose of IMP or currently ≥grade 2 bleeding or factors judged by the investigator to have a high risk of bleeding (such as active peptic ulcer or esophageal varices) at present;
* The adverse reactions of previous anti-tumour treatments have not yet recovered to CTCAE 5.0 grade evaluation ≤1 (except for toxicity judged by the investigator to have no safety risk, such as hair loss, grade 2 peripheral neurotoxicity, etc.);
* Central nervous system metastasis or meningeal metastasis with clinical symptoms, or other evidence that the subject's central nervous system metastasis or meningeal metastasis has not been controlled, and the investigator judges it to be unsuitable for inclusion;
* Gastrointestinal perforation, abdominal fistula, or intra-abdominal abscess occurred within 6 months before the first dose of the IMP; or the investigator has determined that there are high-risk factors for the formation of cavity organ perforation/fistula (such as tumour infiltration in the cavity Outer layer of the wall); inflammatory bowel disease (including ulcerative colitis and Crohn's disease), diverticulitis, cholecystitis, symptomatic cholangitis or appendicitis;
* Unable to be dosed orally, or there are conditions that have been judged by the investigators to seriously affect the absorption of the gastrointestinal tract, such as dysphagia, nausea and vomiting that are difficult to control, intestinal obstruction, and gastric outlet obstruction;
* Have active infection 1 week before the first dose of IMP and currently need systemic anti-infective treatment;
* HIV infection, active HBV infection (HBV DNA exceeds the ULN), active HCV infection (HCV RNA exceeds the ULN);
* Have a history of serious cardiovascular and cerebrovascular diseases, including but not limited to: Severe heart rhythm or conduction abnormalities, such as ventricular arrhythmia that requires clinical intervention, grade Ⅱ-Ⅲ atrioventricular block, etc.; Thromboembolic events requiring therapeutic anticoagulation, or subjects with venous filters;According to the New York Heart Association (NYHA) standards, subjects with grade III~IV cardiac insufficiency;Acute coronary syndrome, congestive heart failure, aortic dissection, stroke or other cardiovascular and cerebrovascular events of grade 3 or above occurred within 6 months before the first administration of IMP;Clinically uncontrollable hypertension (blood pressure cannot be controlled at systolic blood pressure <140 mmHg and diastolic blood pressure <90 mmHg after standard antihypertensive treatment);Any factors that increase the risk of QTc prolongation or arrhythmia, such as heart failure, hypokalemia, congenital long QT syndrome, use of any concomitant drugs that are known or may prolong the QT interval (see Appendix 5 for details);
* The third gap effusion that cannot be controlled clinically is not suitable for inclusion in the study judged by the investigator;
* Known history of drug abuse;
* Subjects with mental disorders or poor compliance;
* Women who are pregnant or breastfeeding;
* Cannot tolerate venous blood sampling;
* Known to be allergic to LM-061 tablets or any of its excipients;
* Has history of other serious systemic diseases judged by the investigator, or other reasons are not suitable for participating in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-05-20 (Actual); Primary Completion 2023-02-07 (Actual); Study Completion 2023-07-19 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events and serious adverse events | From screening up to 1.5 year
  The safety profile of LM061 will be assessed by monitoring the adverse events (AE) per the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) v5.0
Dose-limiting toxicities (DLT) | Cycle 1 of each cohort. Duration of one cycle is 28 days
  DLT is defined as a toxicity (adverse event at least possibly related to LM061) occurring during the DLT observation period (the initial 21 days)
Maximum tolerated dose (MTD) | Cycle 1 of each cohort. Duration of one cycle is 28 days
  MTD is defined as the dose for which the probability of DLT does not exceed the upper bound of the EI, 0.35, and is closest to the target toxicity probability p_T=0.3 during the DLT assessment period (from LM-061 single dose to the first treatment cycle of the multiple dose).
  The i3+3 design does not select a dose as the MTD unless at least 3 subjects have completed the safety assessment.
Change in Vital Signs-ear temperature | Baseline (Week 0) through approximately 1 year after first administration of LM061
  Change in vital signs-ear temperature will be measured after the subject has been fully rested.
Change in Vital Signs-pulse rate | Baseline (Week 0) through approximately 1 year after first administration of LM061
  Change in vital signs-pulse rate will be measured after the subject has been fully rested.
Change in Vital Signs-blood pressure | Baseline (Week 0) through approximately 1 year after first administration of LM061
  Change in vital signs-blood pressure will be measured after the subject has been fully rested.
Change in Electrocardiogram (ECG)-RR interval | Baseline (Week 0) through approximately 1 year after first administration of LM061
  RR interval of 12-lead ECG will be performed in the supine position after the patients are fully rested at each timepoint for once. RR is the standard heart rate which calculated by 60 divided by heart rate.
Change in Electrocardiogram (ECG)-QT interval | Baseline (Week 0) through approximately 1 year after first administration of LM061
  QT interval of 12-lead ECG will be performed in the supine position after the patients are fully rested at each timepoint for once.
Change in Electrocardiogram (ECG)-QRS duration | Baseline (Week 0) through approximately 1 year after first administration of LM061
  QRS duration of 12-lead ECG will be performed in the supine position after the patients are fully rested at each timepoint for once.
Incidence of Abnormal Clinical Laboratory Test Results-hematology | Baseline (Week 0) through approximately 1 year after first administration of LM061
  Number of participants with incidence of abnormal clinical lab test results like hematology will be assessed.
Incidence of Abnormal Clinical Laboratory Test Results-Biochemistry | Baseline (Week 0) through approximately 1 year after first administration of LM061
  Number of participants with incidence of abnormal clinical lab test results like Biochemistry will be assessed.
Incidence of Abnormal Clinical Laboratory Test Results-Urinalysis | Baseline (Week 0) through approximately 1 year after first administration of LM061
  Number of participants with incidence of abnormal clinical lab test results like Urinalysis will be assessed.
Incidence of Abnormal Clinical Laboratory Test Results-Coagulation test | Baseline (Week 0) through approximately 1 year after first administration of LM061
  Number of participants with incidence of abnormal clinical lab test results like Coagulation test will be assessed.

SECONDARY OUTCOMES:
Area under the serum concentration versus time curve within one dosing interval (AUCtau) | Up to 1.5year
  To determine the pharmacokinetics (PK) profile of LM061 Single dose: pre-dose (within 30 minutes before administration), and 1 h, 3 h, 6 h, 8 h, 10 h, 12 h, 24 h, 36 h, 48 h, 72 h, 96 h after administration on C0D1; Multiple dose: pre-dose (within 30 minutes before administration) on C1D1, C1D8, and C1D15; pre-dose (within 30 minutes before administration), and 1 h, 3 h, 6 h, 8 h, 10 h, 12 h, 24 h after administration on C1D22;
  The timepoints of PK sample may be adjusted base on the human PK data. The blood samples for PK analysis will be collected as much as possible if the subjects end of treatment/early withdraw.
Volume of distribution (Vd) | Up to 1.5 year
  To determine the pharmacokinetics (PK) profile of LM061 For AML, the efficacy will be evaluated by using the European LeukemiaNet (ELN) 2017 criteria. The complete blood count and bone marrow will be evaluated at screening visit and every 4 weeks ± 1 week (relative to C1D1) after the start of multiple administrations until the progressive disease judged by investigator or initiate new anti-tumour therapy or subject withdraw. The assessment results are divided into complete remission (CR), CR without minimal residual disease (CRMRD-)，CR with incomplete hematologic recovery (CRi), morphologic leukemia-free state (MFLS), partial remission (PR), stable disease (SD), progressive disease (PD).
Volume of distribution at steady state (Vss) | Up to 1.5 year
  To determine the pharmacokinetics (PK) profile of LM061
Maximum serum concentration (Cmax) | Up to 1.5 year
  To determine the pharmacokinetics (PK) profile of LM061
Trough concentration before the next dose is administered (Ctrough) | Up to 1.5year
  To determine the pharmacokinetics (PK) profile of LM061
Time to reach maximum serum concentration (Tmax) | Up to 1.5 year
  To determine the pharmacokinetics (PK) profile of LM061
Clearance (CL) | Up to 1.5 year
  To determine the pharmacokinetics (PK) profile of LM061
Terminal half-life (T1/2) | Up to 1.5 year
  To determine the pharmacokinetics (PK) profile of LM061
Dose proportionality | Up to 1.5 year
  To determine the pharmacokinetics (PK) profile of LM061
Objective response rate (ORR) | Up to 1.5 year
  To assess the preliminary antitumor activity of LM102,The ORR, using RECIST 1.1 criteria, was defined as the percentage of participants in the analysis population who had a confirmed Complete Response (CR; disappearance of all target lesions) or Partial Response (PR; at least a 30% decrease in the sum of diameters of target lesions) at any time during the study, based on Investigator assessment.
Best of response (BOR) | Up to 1.5 year
  To assess the preliminary antitumor activity of LM061
Disease control rate (DCR) | Up to 1.5 year
  To assess the preliminary antitumor activity of LM061

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai City, China

IPD SHARING:
Plan to Share IPD: No